CLINICAL TRIAL: NCT01193855
Title: Single Site, Phase II, Double Blind, Randomized, Placebo Controlled Study of the Effect of Dutasteride (Avodart) 0.5mg on the Volume and Characteristics of Prostate Cancer, as Assessed by Multifunctional Magnetic Resonance Imaging (MRI) With Lower Risk Prostate Cancer Suitable for Active Surveillance. (MAPPED TRIAL)
Brief Title: Dutasteride in Treating Patients With Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College London Hospitals (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000684018; UCL-09-0221; EUDRACT-2009-012405-18; EU-21067
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Prostate Cancer
Keywords: stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dutasteride; Watchful Waiting; High-Energy Shock Waves

INTERVENTIONS:
Drug: dutasteride
Drug: gadolinium-chelate
Other: active surveillance
Procedure: diffusion-weighted magnetic resonance imaging
Procedure: functional magnetic resonance imaging
Procedure: prostate biopsy
Procedure: ultrasound imaging

SUMMARY:
RATIONALE: Dutasteride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This randomized phase II trial is studying how well giving dutasteride works in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the change in volume of foci of prostate cancer as assessed by T2-weighted MRI, following exposure to dutasteride (Avodart) 0.5 mg daily for six months.

Secondary

* To determine the change in volume of prostate cancer as determined by gadolinium-enhanced MRI and diffusion-weighted MRI after 6 months of dutasteride 0.5 mg compared to placebo.
* To determine the change in volume of prostate cancer as determined by T2-weighted MRI, gadolinium-enhanced MRI, and diffusion-weighted MRI after 3 months of dutasteride compared to placebo.
* To determine the changes in MR characteristics of prostate cancer (perfusion, cell density) between baseline and six months in patients on dutasteride compared to placebo.
* To determine the change in volume of prostate cancer as assessed by HistoScan transrectal ultrasound between baseline and six months, in patients on dutasteride compared to placebo.
* To determine the association between the measured prostate cancer volumes on MRI with the measured prostate cancer volumes on HistoScan at baseline and six months in patients on dutasteride compared to placebo.
* To determine the association between the measured changes in prostate cancer volume using MRI, and the measured changes in prostate cancer volume using HistoScan transrectal ultrasound, at baseline and at six months, in patients on dutasteride compared to placebo.
* To correlate changes in tumor volume and characteristics seen on MRI with changes seen on HistoScan between baseline and six months in patients on dutasteride compared to placebo.
* To correlate change in tumor volume and characteristics seen on MRI with histological features as seen on 6-month biopsy (Gleason score and sum, number of cores involved, cancer core length) in patients on dutasteride compared to placebo.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral dutasteride once daily for 6 months. Treatment continues in the absence of unacceptable toxicity.
* Arm II: Patients receive oral placebo once daily for 6 months. Treatment continues in the absence of unacceptable toxicity.

Patients undergo a multi-sequence MRI at baseline, 3 months, and 6 months and HistoScan transrectal ultrasound at baseline and 6 months. Patients may also undergo a targeted biopsy of the prostate (standard transrectal biopsy plus ultrasound-guided targeting of lesions seen on MRI) at 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer, meeting all of the following criteria:

  * Prostate-specific antigen (PSA) < 10.0 ng/mL
  * T1c-T2a disease
  * Gleason sum of 6 or 7 (secondary pattern 4 only)
* Patients with low risk disease must meet the following criteria:

  * Gleason pattern 3 + 3
  * PSA < 10.0 ng/mL
  * Clinical T2a disease
* Patients with Gleason secondary pattern 4 (i.e., Gleason Pattern 3 + 4) are eligible but must not have a primary pattern 4, PSA > 10 ng/mL, or clinical T2b disease
* Measurable disease on MRI of at least 0.2 cc, based on planimetry volume
* Biopsy-proven disease within 2 years of screening visit

  * No biopsy artifact on MRI scan (minimum 12-week interval between biopsy and baseline MRI)
* Eligible for active surveillance according to the criteria set out by the National Institute for Health and Clinical Excellence

PATIENT CHARACTERISTICS:

* ALT and AST ≤ 2 times the upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2 times ULN
* Bilirubin ≤ 1.5 times ULN
* Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min
* Able to swallow and retain oral medication
* Able and willing to participate in the study for its duration
* Able to read and write (health-outcomes questionnaires are written)
* Able to understand instructions related to study procedures and give written informed consent
* No history of another malignancy within five years that could affect the diagnosis of prostate cancer
* No history or current evidence of drug or alcohol abuse within the last 12 months that might confound the results of the study or pose additional risk to the patient
* No known hypersensitivity to any 5α-reductase inhibitor or to any drug chemically related to dutasteride
* No contraindication for undergoing gadolinium-enhanced MRI, including any of the following:

  * Inability to see tumor focus of ≥ 0.2 cc on T2 sequences
  * Previous allergic reaction to gadolinium
  * Serum creatinine > ULN
  * Incompatible pacemaker
  * Metal fragments in eyes
  * Hip replacements that give artifact with prostate/pelvis views
  * Any artifact or condition that reduces image quality of MRI (e.g., inability to keep still)
* No unstable serious co-existing medical condition(s) including, but not limited, to any of the following:

  * Myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident within 6 months prior to screening visit
  * Uncontrolled diabetes
  * Peptic ulcer disease uncontrolled by medical management

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy (external-beam or brachytherapy), high-intensity focused ultrasound (HIFU), or photodynamic therapy (PDT)
* No prior chemotherapy
* At least 3 months since prior and no concurrent prostatic surgery, including TUNA, TURP, TUIP, laser treatment, thermotherapy, balloon dilatation, prosthesis, and ultrasound ablation
* No prior oral glucocorticoids

  * Glucocorticoids, except inhaled or topical, are not permitted within 3 months prior to visit one
* No prior GnRH analogues (e.g., leuprolide, goserelin)
* No prior or concurrent hormonal treatment (e.g., megestrol, medroxyprogesterone, cyproterone, DES) of prostate cancer
* No current and/or prior use of the following medications:

  * Finasteride (Proscar, Propecia), or dutasteride (GI198745, AVODART) exposure within 12 months prior to study entry
  * Any other investigational 5α-reductase inhibitors within the past 12 months
  * Anabolic steroids within the past 6 months
  * Drugs with antiandrogenic properties within the past 6 months (e.g., spironolactone, flutamide, bicalutamide, cimetidine, ketoconazole, progestational agents)

    * The use of cimetidine is permitted prior to study entry
    * The use of topical ketoconazole is permitted prior to and during the study
* No participation in another investigational or marketed drug trial within the 30 days prior to the first dose of study drug or anytime during the study period

Max Age: 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
The change in volume of foci of prostate cancer (PC) as assessed by T2-weighted (T2w) MRI between baseline and 6 months

SECONDARY OUTCOMES:
The change in volume of PC as determined by gadolinium-enhanced (GE) MRI and diffusion-weighted (DW) MRI at 6 months
The change in volume of PC as determined by T2w MRI, GE MRI, and DW MRI at 3 months
The changes in MR characteristics of PC (perfusion, cell density) between baseline and 6 months
The change in volume of PC as assessed by HistoScan transrectal ultrasound (TRUS) between baseline and 6 months
The association between the measured PC volumes on MRI with the measured PC volumes on TRUS at baseline and 6 months
The association between the measured changes in PC volume using MRI vs TRUS at baseline and 6 months
The association of PC volume change with qualitative changes seen on TRUS between baseline and 6 months
The association between MR changes in volume and characteristics with histological features as seen on 6-month biopsy (Gleason score and sum, number of cores involved, cancer core length)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Emberton, MD, FRCS, MBBS, Principal Investigator — University College London Hospitals
Locations (1):
- University College of London Hospitals, London, England, United Kingdom